CLINICAL TRIAL: NCT07323212
Title: Occupational Impacts of Compound Resistance Training in Community-Dwelling Older Adults
Brief Title: Occupational Impacts of Resistance Training in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Washington Regional Medical Center (Other)
Responsible Party: Principal Investigator, Alexis R. Skalberg, Principal Investigator, University of Arkansas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 298900
Record Dates: First submitted 2025-12-03; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Resistance Training; Older Adults (65 Years and Older)

STUDY DESIGN:
Intervention Model Description: Quasi-experimental pre-test post-test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants engaged in intervention
  Interventions: Other: Compound Resistance Training

INTERVENTIONS:
Other: Compound Resistance Training — Intervention will take place over the course of 10 weeks, with individual sessions occurring twice weekly for one hour per session with each participant. Each session will consist of personalized strength training sessions, utilizing programming with a focus on compound, multi-joint movements, in keeping with existing literature on the subject.

SUMMARY:
This study aims to assess the impact of compound resistance training on the ability of adults age 65 and older to participate in desired daily activities, their satisfaction with their level of participation, and their overall mental health.

DETAILED DESCRIPTION:
Eligible and consented participants will complete pre-assessment questionnaires: the Patient Health Questionnaire-9, the Perceived Stress Scale-10, and the Canadian Occupational Performance Measure. Participants will also engaged in a semi-structured interview with pre-set questions. Following pre-assessment, all data will be coded and stored in encrypted software through the university. Participants will then engage in a 10-week intervention period consisting of two 1-hour sessions strength training with principal investigator guiding participants for safety, form, intensity, and volume of exercises. Modifications will be made to exercise programming based on individual performance and individual needs, in accordance with occupational therapy best practices. Rate of Perceived Exertion (RPE) will be used as a guide for intensity with the aim being self-reported RPE 7-8 for each exercise. At completion of the intervention period, participants will complete post-assessment questionnaires: the Patient Health Questionnaire-9, the Perceived Stress Scale-10, and the Canadian Occupational Performance Measure. Participants will also engaged in another semi-structured interview with pre-set questions. Data will be analyzed for statistical and clinically significant changes.

ELIGIBILITY:
Inclusion Criteria:

* Adult age 65 or older

  * Living independently in a community dwelling, such as a house or apartment
  * Able to complete basic daily tasks (i.e. dressing, toileting, transfers) without assistance from another person
  * Access to transportation to and from sessions for this study
  * Able to attend two, one-hour sessions per week for the duration of the study
  * Has a membership to Silver Sneakers, Silver and Fit, and/or Renew Active, or are willing to obtain a paid membership to Washington Regional Center for Exercise

Exclusion Criteria:

* · Personal history of stroke or heart attack

  * Limb amputation
  * Heart failure or arrythmias
  * Presence of brain or aortic aneurism
  * Active cancer
  * Major illness
  * Physical activity contraindicated as instructed by a physician
  * Active drug abuse
  * Moderate to severe cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | Baseline and 10 weeks
  Occupational therapy questionnaire
  Section 1: Performance Participants requested to report their perception of their performance of a given occupation/activity/daily task on a scale of 1 to 10, with 1 being "unable to do it at all" and 10 being "able to do it with no issues at all".
  Section 2: Satisfaction Participants requested to reported their satisfaction with their currently level of performance with the previously reported occupation/activity/daily task on a scale of 1 to 10, with 1 being "completely dissatisfied" and 10 being "completely satisfied".
  Higher scores on either or both sections indicate a better outcome.
Patient Health Questionnaire-9 | Baseline and 10 weeks
  Mental health questionnaire (depression screen)
  Participants asked to report the frequency of depression symptoms listed on form over the last 2 weeks using a scale from 0 to 3. Reporting 0 indicates "not at all", reporting 1 indicates "several days", reporting 2 indicates "more than half the days", reporting 3 indicates "nearly every day". Lower scores indicate a better outcome
Perceived Stress Scale-10 | Baseline and 10 weeks
  Mental health questionnaire (stress screen)
  Participants asked to report frequency of stress impacts on daily life by responding how many days in the past month the participant felt or thought a certain way. Answers are on a scale of 0-4. Reporting 0 indicates "never", reporting 1 indicates "almost never", reporting 2 indicates "sometimes", reporting 3 indicates "fairly often", and reporting 4 indicates "very often". Lower scores indicate better results.
Reported perceptions of exercise, self-confidence, and confidence in gym environment | baseline and 10 weeks
  Qualitative data: word associations, open responses, takeaways from study. Thematic analysis and coding for frequency of themes

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Muriithi, OTD, Study Chair — University of Arkansas
Locations (1):
- Washington Regional Center for Exercise, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD (coded)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start date 12/3/2025 end date 12/3/2030 or at time of acceptance for publication, whichever comes first
Access Criteria: Dr. Jennifer Muriithi, faculty capstone mentor at university where student is affiliated

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT07323212/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT07323212/ICF_001.pdf